CLINICAL TRIAL: NCT06964620
Title: Efficacy and Safety of Sanggua Tablets in the Treatment of Patients With Impaired Glucose Tolerance and Mild Type 2 Diabetes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Gang Yuan, Principal Investigator, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20241010
Record Dates: First submitted 2025-04-12; First posted 2025-05-09 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; Impaired Glucose Tolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional treatment plus Sanggua tablets (Experimental): Conventional treatment plus Sanggua tablets (0.75 g per tablet, twice daily, bid) for 16 weeks
  Interventions: Drug: Sanggua tablets
- Conventional treatment plus placebo (Placebo Comparator): Conventional treatment plus placebo (0.75 g per tablet, twice daily, bid) for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sanggua tablets — Patients will continue their background medications and receive Sang Gua tablets, twice daily (bid).
  Arms: Conventional treatment plus Sanggua tablets
Drug: Placebo — Patients will continue their background medications and receive placebo, twice daily (bid).
  Arms: Conventional treatment plus placebo

SUMMARY:
Type 2 diabetes mellitus (T2DM) and impaired glucose tolerance (IGT) are growing public health challenges. Early intervention in mild T2DM and IGT is essential to prevent disease progression and severe complications. Traditional Chinese Medicine (TCM) provides a potential therapeutic approach.

Sanggua tablets, a TCM formula composed of mulberry leaf, bitter melon, kudzu root, Chinese yam, and cassia seed, embody TCM principles of clearing heat, generating body fluids, tonifying the spleen and stomach, and nourishing the lungs and kidneys. Modern studies show that Sanggua tablets effectively lower blood glucose and improve lipid profiles through components like mulberry polysaccharides and bitter melon saponins. These findings suggest their potential as an alternative or complementary therapy for mild T2DM and IGT.

This study will conduct a randomized, double-blind, placebo-controlled, parallel-group clinical trial among patients with IGT and mild T2DM. Participants will receive a 16-week intervention with Sanggua tablets. The primary outcome is glycated hemoglobin (HbA1c), with secondary outcomes such as fasting blood glucose (FBG), fasting insulin (FINS), HOMA-IR, lipid profiles and so on. Safety will be closely monitored. Additionally, fecal samples will be collected for 16S rDNA sequencing to explore the role of gut microbiota in the therapeutic effects of Sanggua tablets. This study aims to provide evidence for the clinical application and development of Sanggua tablets as a novel TCM therapy.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) and impaired glucose tolerance (IGT) are significant public health concerns, with rising prevalence rates globally. Treating mild T2DM and IGT is crucial to prevent disease progression and reduce the risk of severe complications such as cardiovascular diseases. Traditional Chinese Medicine (TCM) offers a promising approach in this context.

Sanggua tablets, a TCM formula, consist of mulberry leaf, bitter melon, kudzu root, Chinese yam, and cassia seed. These ingredients work synergistically to achieve the TCM therapeutic principles of clearing heat and detoxifying, generating body fluids and moistening dryness, tonifying the spleen and stomach, and nourishing the lungs and kidneys. Modern pharmacological studies have shown that Sanggua tablets have significant therapeutic potential. Their components, such as mulberry polysaccharides and bitter melon saponins, have been proven to lower blood glucose levels by promoting glycogen synthesis and inhibiting glucose absorption. Additionally, they have demonstrated hypolipidemic effects, improving lipid profiles and potentially preventing atherosclerosis.

Clinical and experimental evidence suggests that Sanggua tablets can effectively improve insulin resistance and regulate lipid metabolism. These findings highlight their potential as an alternative or complementary therapy for mild T2DM and IGT. Further research is needed to elucidate their mechanisms of action and optimize their clinical application.

This study proposes to employ a randomized, double-blind, placebo-controlled, parallel-group clinical trial design. The study population will consist of patients with IGT and mild T2DM. Participants will undergo a 16-week intervention with Sanggua tablets. The primary outcome is glycated hemoglobin (HbA1c), with secondary outcomes such as fasting blood glucose (FBG), fasting insulin (FINS), HOMA-IR, lipid profiles and so on. Safety indicators will also be closely monitored. The clinical efficacy of Sanggua tablets will be re-evaluated through these measures. Additionally, to explore its mechanism of action, fecal samples will be collected from participants for 16S rDNA sequencing to investigate the role of gut microbiota. This study aims to provide evidence for the clinical application and potential development of Sang Gua tablets as a Category 1.1 innovative traditional Chinese medicine.

Based on calculations using the PASS 15 software, a total of 84 participants are required for enrollment, with 42 participants in each group.

Initially screened participants will undergo baseline assessments during the screening period (V0, from Day -7 to Day 0) to determine their eligibility based on the inclusion and exclusion criteria. Randomization of eligible participants and the preparation of randomization envelopes will follow the principles of randomized clinical trial design. Participants meeting the inclusion and exclusion criteria will be randomly assigned to two groups in a 1:1 ratio, receiving either conventional treatment plus Sanggua tablets or conventional treatment plus placebo. Both Sanggua tablets and the placebo will be manufactured by Wuhan Jianmin Dapeng Pharmaceutical Co., Ltd. Random numbers generated using SAS software will be used to determine the codes for participants in the two groups. Two copies of the randomization envelopes will be prepared, sealed, and separately stored by the investigator and the person in charge of the clinical study. After 16 weeks of treatment, the efficacy and safety of the interventions will be evaluated.

Study Visits:

V0 (Screening): Conducted 7 days before enrollment, includes assessments such as physical examination, vital signs, fasting blood glucose (FBG), glycated hemoglobin (HbA1c).

V1 (Enrollment): Occurs on Day 0, where participants are assigned to groups and begin treatment.

V2 (4 weeks): Participants are assessed for FBG, vital signs, and other routine checks.

V3 (8 weeks): Participants are assessed for FBG, vital signs, and additional assessments.

V4 (12 weeks): Participants are assessed for FBG and vital signs assessment. V5 (16 weeks): Final assessment includes physical examination, vital signs, FBG, HbA1c, oral glucose tolerance test (OGTT), and other glycemic and lipid profiles.

V6 (Post-study): Follow-up 28 days after the last dose, includes a telephone interview for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with impaired glucose tolerance (IGT).
* Patients aged 18-70 diagnosed with type 2 diabetes mellitus (T2DM) deemed by the clinician not requiring pharmacological intervention.
* Glycated hemoglobin (HbA1c) levels between 5.6% and 7.5%.
* Voluntarily sign an informed consent form before the commencement of trial-related activities, understand the procedures and methods of the trial, and are willing and able to strictly adhere to the clinical trial protocol to complete the study.

Exclusion Criteria:

* Type 1 diabetes mellitus.
* Known allergies to Sang Gua tablets or any of its components.
* Use of hypoglycemic or lipid-lowering drugs within the last three months.
* Presence of severe primary or secondary respiratory, cardiovascular, hepatic, or renal diseases, rheumatic connective tissue diseases, or hematological disorders.
* Uncontrolled or unstable conditions exacerbated by infections, severe electrolyte imbalances, or other factors.
* Patients with primary or secondary kidney diseases, hypertension, heart failure, acidosis, or urinary tract infections causing increased urinary protein, excepted.
* Patients with psychiatric disorders.
* Pregnant or planning to become pregnant women, or nursing mothers.
* Patients requiring long-term steroid therapy.
* Patients with poorly controlled hypertension or secondary hypertension.
* Patients who have participated in other clinical trials within the past three months.
* Patients deemed by the investigator as unsuitable for this clinical trial due to potential interference with trial results, impediments to full participation in the study, medical history, disease evidence, abnormal treatments, or laboratory values, or any other condition considered by the investigator to pose potential risks for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-22 (Estimated); Primary Completion 2027-11-24 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c, %) | The percentage of glycated hemoglobin will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  The percentage of glycated hemoglobin in the blood will be determined to evaluate the hypoglycemic effect of Sanggua tablets. Evaluate the degree of reduction in glycated hemoglobin after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.

SECONDARY OUTCOMES:
Fasting blood glucose (FBG, mmol/L) | FBG will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), Week 8 (V3), Week 12 (V4), and Week 16 (V5).
  Fasting blood glucose is the concentration of glucose in the blood after an overnight fast, assessing the effectiveness of Sang Gua tablets on lowering blood glucose. Evaluate the degree of reduction in FBG after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
2 hour blood glucose (mmol/L) | FBG will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), Week 8 (V3), Week 12 (V4), and Week 16 (V5).
  The oral glucose tolerance test (OGTT) involves fasting, consuming a glucose-rich drink, containing 75 grams of glucose, and having blood glucose levels measured 2 hours later to assess how well the body processes glucose, testing the tablets' ability to manage glucose metabolism. 2 hour blood glucose is the concentration of glucose in the blood after OGTT 2h, assessing the effectiveness of Sang Gua tablets on lowering blood glucose. Evaluate the degree of reduction in 2 hour glucose after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Fasting insulin (FINS, uIU/ml) | FINS will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  The oral glucose tolerance test (OGTT) involves fasting, consuming a glucose-rich drink, containing 75 grams of glucose, and having blood insuiin levels measured at the begining, testing the tablets' ability to manage glucose metabolism. Fasting insulin is the concentration of insulin in the blood after an overnight fast, evaluating the tablets' impact on insulin secretion. Evaluate the degree of reduction in FINS after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
2 hour insulin (uIU/ml) | FINS will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  The oral glucose tolerance test (OGTT) involves fasting, consuming a glucose-rich drink, containing 75 grams of glucose, and having blood insulin levels measured 2 hours later, testing the tablets' ability to manage glucose metabolism. 2 hour insulin is the concentration of insulin in the blood after OGTT 2h, evaluating the tablets' impact on Insulin resistance. Evaluate the degree of reduction in 2 hour insulin after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Fasting C-peptide(ug/L) | C-peptide will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  The oral glucose tolerance test (OGTT) involves fasting, consuming a glucose-rich drink, containing 75 grams of glucose, and having C-peptide levels measured at the begining. Fasting C-peptide is the concentration of C-peptide in the blood after an overnight fast, indicating the tablets' effect on pancreatic function. Evaluate the degree of reduction in fasting C-peptide after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
2 hour C-peptide(ug/L) | C-peptide will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  The oral glucose tolerance test (OGTT) involves fasting, consuming a glucose-rich drink, containing 75 grams of glucose, and having C-peptide levels measured 2 hours later. 2 hour C-peptide is the concentration of C-peptide in the blood after OGTT 2h, indicating the tablets' effect on pancreatic function. Evaluate the degree of reduction in 2 hour C-peptide after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Homeostasis model assessment of insulin resistance (HOMA-IR) | HOMA-IR will be calculated at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  The Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) is calculated as fasting insulin (uU/L)×fasting glucose (mmol/L)/22.5, determining the tablets' influence on insulin sensitivity. Evaluate the degree of reduction in HOMA-IR after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
HOMA-β | HOMA-β will be calculated at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  HOMA-β is calculated as 20×fasting insulin (mU/L)/(fasting glucose (mmol/L)-3.5), which estimates the tablets' effect on beta-cell function. Evaluate the degree of rise in HOMA-β after the end of the treatment period of the patients and the rate of rise among the 84 enrolled patients.
TAR (Time Above Range > 13.9 mmol/L) | Participants will wear CGM devices for two weeks starting one week prior to enrollment, and again for two weeks at the end of the treatment period, beginning one week before the final medication administration.
  Monitoring Continuous Glucose Monitoring (CGM) metrics is crucial for assessing Sanggua tablets's impact on glucose control, identifying fluctuations, and evaluating the overall effectiveness and safety of the treatment in managing blood sugar levels. TAR (Time Above Range > 13.9 mmol/L) indicates the proportion of time with severe hyperglycemia, suggesting a high risk. Evaluate the degree of change of TAR (Time Above Range > 13.9 mmol/L) after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
TAR (Time Above Range 10.1-13.9 mmol/L) | Participants will wear CGM devices for two weeks starting one week prior to enrollment, and again for two weeks at the end of the treatment period, beginning one week before the final medication administration.
  Monitoring Continuous Glucose Monitoring (CGM) metrics is crucial for assessing Sanggua tablets's impact on glucose control, identifying fluctuations, and evaluating the overall effectiveness and safety of the treatment in managing blood sugar levels. TAR (Time Above Range 10.1-13.9 mmol/L) indicates the proportion of time with moderate hyperglycemia. Evaluate the degree of change of TAR (Time Above Range 10.1-13.9 mmol/L) after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
TIR (Time in Range 3.9-10.0 mmol/L) | Participants will wear CGM devices for two weeks starting one week prior to enrollment, and again for two weeks at the end of the treatment period, beginning one week before the final medication administration.
  Monitoring Continuous Glucose Monitoring (CGM) metrics is crucial for assessing Sanggua tablets's impact on glucose control, identifying fluctuations, and evaluating the overall effectiveness and safety of the treatment in managing blood sugar levels. TIR (Time in Range 3.9-10.0 mmol/L) represents the proportion of time blood glucose levels are within the target range. Evaluate the degree of change of TIR (Time in Range 3.9-10.0 mmol/L) after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
TBR (Time Below Range 3.0-3.8 mmol/L) | Participants will wear CGM devices for two weeks starting one week prior to enrollment, and again for two weeks at the end of the treatment period, beginning one week before the final medication administration.
  Monitoring Continuous Glucose Monitoring (CGM) metrics is crucial for assessing Sanggua tablets's impact on glucose control, identifying fluctuations, and evaluating the overall effectiveness and safety of the treatment in managing blood sugar levels. TBR (Time Below Range 3.0-3.8 mmol/L) indicates the proportion of time with mild hypoglycemia. Evaluate the degree of change of TBR (Time Below Range 3.0-3.8 mmol/L) after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
TBR (Time Below Range <3.0 mmol/L) | Participants will wear CGM devices for two weeks starting one week prior to enrollment, and again for two weeks at the end of the treatment period, beginning one week before the final medication administration.
  Monitoring Continuous Glucose Monitoring (CGM) metrics is crucial for assessing Sanggua tablets's impact on glucose control, identifying fluctuations, and evaluating the overall effectiveness and safety of the treatment in managing blood sugar levels. TBR (Time Below Range <3.0 mmol/L) indicates the proportion of time with severe hypoglycemia, suggesting a low risk. Evaluate the degree of change of TBR (Time Below Range <3.0 mmol/L) after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
Coefficient of variation | Participants will wear CGM devices for two weeks starting one week prior to enrollment, and again for two weeks at the end of the treatment period, beginning one week before the final medication administration.
  Monitoring Continuous Glucose Monitoring (CGM) metrics is crucial for assessing Sanggua tablets's impact on glucose control, identifying fluctuations, and evaluating the overall effectiveness and safety of the treatment in managing blood sugar levels. Glucose Fluctuations will be assessed using the coefficient of variation (CV) to reflect the stability of blood glucose levels. Evaluate the degree of change of Coefficient of variation after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
Mean sensor glucose | Participants will wear CGM devices for two weeks starting one week prior to enrollment, and again for two weeks at the end of the treatment period, beginning one week before the final medication administration.
  Monitoring Continuous Glucose Monitoring (CGM) metrics is crucial for assessing Sanggua tablets's impact on glucose control, identifying fluctuations, and evaluating the overall effectiveness and safety of the treatment in managing blood sugar levels. Mean sensor glucose provides an overall assessment of blood glucose levels. Evaluate the degree of change of Mean sensor glucose after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
Glucose Management Index (GMI) | Participants will wear CGM devices for two weeks starting one week prior to enrollment, and again for two weeks at the end of the treatment period, beginning one week before the final medication administration.
  Monitoring Continuous Glucose Monitoring (CGM) metrics is crucial for assessing Sanggua tablets's impact on glucose control, identifying fluctuations, and evaluating the overall effectiveness and safety of the treatment in managing blood sugar levels. Glucose Management Index (GMI) evaluates the long-term effectiveness of blood glucose control. Evaluate the degree of change of Glucose Management Index (GMI) after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
Total Cholesterol（TC,mmol/L） | TC will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Total Cholesterol will be assessed to determine the impact of Sanggua tablets on overall cholesterol levels, providing insight into its lipid-lowering efficacy. Evaluate the degree of reduction in TC after the end of the treatment period of the patients and the rate of rise among the 84 enrolled patients.
Triglycerides（TG, mmol/L） | TG will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Triglycerides will be measured to evaluate the effect of Sanggua tablets on reducing triglyceride levels, a key marker of dyslipidemia and cardiovascular risk. Evaluate the degree of reduction in TG after the end of the treatment period of the patients and the rate of rise among the 84 enrolled patients.
Low-density lipoprotein cholesterol（LDL-C, mmol/L） | LDL-C will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Low-density lipoprotein cholesterol wil be monitored to evaluate Sanggua tablets's ability to lower cholesterol levels, which is crucial for reducing the risk of atherosclerosis and cardiovascular events.. Evaluate the degree of reduction in LDL-C after the end of the treatment period of the patients and the rate of rise among the 84 enrolled patients.
High-density lipoprotein cholesterol（HDL-C, mmol/L） | HDL-C will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  High-density lipoprotein cholesterol will be measured to assess whether Sanggua tablets can increase "good" cholesterol levels, which may enhance cardiovascular protection. Evaluate the degree of rise in HDL-C after the end of the treatment period of the patients and the rate of rise among the 84 enrolled patients.
Lipoprotein(a)（Lp(a), mg/L） | LP(a) will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Lipoprotein(a) will be evaluated to determine Sanggua tablets's effect on this specific lipid marker associated with increased cardiovascular risk, providing a comprehensive assessment of its lipid-modulating properties. Evaluate the degree of reduction in LP(a) after the end of the treatment period of the patients and the rate of rise among the 84 enrolled patients.
Liver Stiffness Measurement(LSM, kPa) | Liver Stiffness Measurement will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Liver transient elastography is a non-invasive procedure that assesses liver stiffness and steatosis by sending shear waves through the liver tissue, which helps in the diagnosis of liver fibrosis and fatty liver disease. A non-invasive test to assess liver health, indicating the tablets' potential effects on liver function. Liver Stiffness Measurement(LSM, kPa) will be examined to evaluate the liver stiffness. Evaluate the degree of reduction in LSM after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Controlled attenuation parameter(CAP, dB/m) | Controlled attenuation parameter will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Liver transient elastography is a non-invasive procedure that assesses liver stiffness and steatosis by sending shear waves through the liver tissue, which helps in the diagnosis of liver fibrosis and fatty liver disease. A non-invasive test to assess liver health, indicating the tablets' potential effects on liver function. Controlled attenuation parameter(CAP, dB/m) will be examined to evaluate steatosis. Evaluate the degree of reduction in CAP after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
C-reactive protein (CRP, mg/L) | CRP will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  C-reactive protein (CRP) is a blood test marker that indicates inflammation in the body, measured to evaluate the tablets' impact on inflammatory processes. Evaluate the degree of reduction in CRP after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Homocysteine(umol/L) | Homocysteine will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Homocysteine is an amino acid whose elevated levels in the blood may indicate an increased risk for cardiovascular disease and is used as a marker for assessing nutritional status and metabolic health. Evaluate the degree of reduction in Homocysteine after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Waist circumference(cm) | Waist circumference will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Measures abdominal fat, assessing the tablets' effect on central obesity, will be used to assess abdominal obesity and related health risks. Evaluate the degree of reduction in waist circumference after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Hip circumference(cm) | Waist circumference will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Measure the hip circumference and evaluate the effect of the tablet on fat distribution, will be used to assess overall obesity and metabolism-related health risks. Evaluate the degree of reduction in hip circumference after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Waist-to-hip ratio | Waist-to-hip ratio will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Waist-to-hip ratio will be used to assess the characteristics of fat distribution, reflect the degree of abdominal fat accumulation, and help determine the regulatory effect of Sanggua tablets on fat distribution. Evaluate the degree of reduction in waist-to-hip ratio after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Waist-to-height ratio | Waist-to-height ratio will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  A simple measure of body proportions, assessing Sanggua tablets' impact on overall body size. Evaluate the degree of reduction in waist-to-height ratio after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Visceral Fat Area (VFA, cm²) | Visceral Fat Area will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  The assessment of body composition provides comprehensive insights into Sanggua tablets's effects on various aspects of physical health. Visceral Fat Area will be assessed to determine the effect on abdominal fat, which is a key risk factor for metabolic syndrome and cardiovascular disease. Evaluate the degree of change of Visceral Fat Area after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
Fecal samples for 16S rDNA sequencing | Fecal samples will be collected at baseline (V1) and at the end of the treatment period(Week 16 ,V5) for 16S rDNA sequencing.
  Fecal samples for 16S rDNA sequencing will be collected to analyze gut microbiota, exploring Sanggua tablets' potential to modulate gut health. Detect the diversity of the intestinal flora, the composition of the dominant flora, potential pathogenic bacteria, the functions of beneficial bacteria, the stability of the flora, and the interaction between the flora and the host. Evaluate the degree of change of each index of fecal samples for 16S rDNA sequencing after the end of the treatment period of the patients and the overall index improvement rate of the 84 enrolled patients.
Body weight(kg) | Body weight will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Body weight monitors changes in weight, assessing the tablets' effect on body mass. Evaluate the degree of reduction in body weight after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Body mass index (BMI) | BMI will be measured at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  Body mass index calculates body fat based on weight and height, evaluating the tablets' impact on body composition. BMI=body weight(kg) / body height(m²). Evaluate the degree of reduction in BMI after the end of the treatment period of the patients and the rate of reduction among the 84 enrolled patients.
Heart rate(time/min) | Heart rate will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), Week 8 (V3), Week 12 (V4), and Week 16 (V5).
  Heart rate monitors heart rate(time/min), assessing the tablets' safety. Evaluate whether these indicators are within the normal range during the treatment period.
Systolic Blood Pressure(mmHg) | Systolic blood pressure will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), Week 8 (V3), Week 12 (V4), and Week 16 (V5).
  Monitoring systolic blood pressure is crucial to ensure that Sanggua tablets treatment does not induce hypertension, a risk factor for cardiovascular events. Evaluate whether systolic blood pressure are within the normal range during the treatment period.
Diastolic Blood Pressure (mmHg) | Diastolic Blood Pressure will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), Week 8 (V3), Week 12 (V4), and Week 16 (V5).
  Assessing diastolic blood pressure is important to verify Sanggua tablets's safety regarding its potential impact on blood pressure regulation and to prevent hypotension-related complications. Evaluate whether diastolic Blood Pressure are within the normal range during the treatment period.
AST(U/L) | AST will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Liver function test evaluates the health of liver, assessing the tablets' safety.The detection of aspartate aminotransferase (AST) levels will be used to assess the potential impact of drugs on liver function, helping to identify whether Sanggua tablets cause liver damage or liver toxicity, thereby ensuring the safety of Sanggua tablets. Evaluate whether these indicators are within the normal range during the treatment period.
ALT(U/L) | ALT will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Liver function test evaluates the health of liver, assessing the tablets' safety. The detection of alanine aminotransferase (ALT) levels will be used to assess the potential impact of drugs on liver function, helping to identify whether Sanggua tablets cause liver damage or liver toxicity, thereby ensuring the safety of Sanggua tablets. Evaluate whether these indicators are within the normal range during the treatment period.
Urea(mmol/L) | Urea will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Kidney function test evaluates the health of kidney, assessing the tablets' safety. The detection of urea levels will be used to assess the impact of Sanggua tablets on renal function and determine whether they interfere with the metabolic and excretory functions of the kidneys, thereby providing an important basis for the safety evaluation of Sanggua tablets. Evaluate whether these indicators are within the normal range during the treatment period.
Blood uric acid(umol/L) | Blood uric acid will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Kidney function test evaluates the health of kidney, assessing the tablets' safety. Detecting uric acid levels will be used to assess the impact of Sanggua tablets on uric acid metabolism in the body and determine whether they may cause or improve the risk of related diseases such as hyperuricemia and gout. Evaluate whether these indicators are within the normal range during the treatment period.
Creatinine(umol/L) | Creatinine will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Kidney function test evaluates the health of kidney, assessing the tablets' safety. The detection of creatinine levels will be used to assess the impact of Sanggua tablets on renal function, to help determine whether the Sanggua tablets have caused renal damage or affected the excretory function of the kidneys. Evaluate whether these indicators are within the normal range during the treatment period.
Bicarbonate(mM) | Bicarbonate will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Kidney function test evaluates the health of kidney, assessing the tablets' safety. The detection of bicarbonate levels will be used to assess the impact of Sanggua tablets on the acid-base balance in the body and determine whether they cause metabolic acidosis or alkalosis, thereby providing an important basis for the safety evaluation of Sanggua tablets. Evaluate whether these indicators are within the normal range during the treatment period.
eGFR(ml/min/1.73m^2) | eGFR will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Kidney function test evaluates the health of kidney, assessing the tablets' safety. The detection and estimation of glomerular filtration rate (eGFR) will be used to assess the impact of Sanggua tablets on renal function, determine whether they have adverse effects on the filtration function of the kidneys, and provide an important basis for the safety evaluation of Sanggua tablets. Evaluate whether these indicators are within the normal range during the treatment period.
ECG PR Interval | ECG PR Interval will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  ECG PR Interval will be used to assess the impact of Sanggua tablets on the atrioventricular conduction system and determine whether there are conduction abnormalities such as atrioventricular block. Evaluate whether these indicators are within the normal range during the treatment period.
ECG QRS Complex | ECG QRS Complex will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  ECG QRS Complex will be used to evaluate the effect of Sanggua tablets on the ventricular depolarization process and determine whether there are ventricular abnormalities such as ventricular hypertrophy and bundle branch block. Evaluate whether these indicators are within the normal range during the treatment period.
ECG QT Interval | ECG QT Interval will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  ECG QT Interval will be used to evaluate the effect of Sanggua tablets on ventricular repolarization, determine whether there is QT interval prolongation, and thereby predict the risk of drug-induced arrhythmias. Evaluate whether these indicators are within the normal range during the treatment period.
ECG P Wave | ECG P Wave will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  ECG P Wave will be used to evaluate the effect of Sanggua tablets on atrial depolarization and determine whether there are atrial abnormalities, such as atrial hypertrophy or atrial fibrillation, etc. Evaluate whether these indicators are within the normal range during the treatment period.
ECG ST Segment | ECG ST Segment will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  ECG ST Segment will be used to evaluate the impact of Sanggua tablets on myocardial ischemia or injury, and to determine whether there is myocardial ischemia, myocardial infarction and other conditions. Evaluate whether these indicators are within the normal range during the treatment period.
ECG T Wave | ECG T Wave will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  ECG T Wave will be used to evaluate the effect of Sanggua tablets on ventricular repolarization and determine whether there are electrolyte disorders or myocardial ischemia and other conditions. Evaluate whether these indicators are within the normal range during the treatment period.
Adverse events and adverse reactions | Adverse events and adverse reactions will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), Week 8 (V3), Week 12 (V4), and Week 16 (V5).
  Monitored to ensure the safety of the tablets and to identify any potential side effects.
White Blood Cell Count (WBC, 10^9/L) | White Blood Cell Count will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Blood routine examination is a standard test that evaluates the levels of red and white blood cells, platelets, and other components in the blood, providing a general overview of health and the tablets' safety. White Blood Cell Count evaluates the impact of Sanggua tablets on the systemic immune function, determine whether there is an infection or inflammatory response, and whether Sanggua tablets causes abnormal increase or decrease in white blood cells. Evaluate whether these indicators are within the normal range during the treatment period.
Absolute Neutrophil Count | Absolute Neutrophil Count will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Blood routine examination is a standard test that evaluates the levels of red and white blood cells, platelets, and other components in the blood, providing a general overview of health and the tablets' safety. Absolute Neutrophil Count detects the effect of Sanggua tablets on neutrophils, determine whether there is neutropenia or increase, and indicate the risk of infection or Sanggua tablets-related bone marrow suppression. Evaluate whether these indicators are within the normal range during the treatment period.
Absolute Lymphocyte Count | Absolute Lymphocyte Count will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Blood routine examination is a standard test that evaluates the levels of red and white blood cells, platelets, and other components in the blood, providing a general overview of health and the tablets' safety. Absolute Lymphocyte Count evaluates the impact of Sanggua tablets on lymphocytes, determine whether there is a decrease or increase in lymphocytes, and indicate changes in immune system function or potential immune-related adverse reactions. Evaluate whether these indicators are within the normal range during the treatment period.
Red Blood Cell Count (RBC, 10^12/L) | Red Blood Cell Count will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Blood routine examination is a standard test that evaluates the levels of red and white blood cells, platelets, and other components in the blood, providing a general overview of health and the tablets' safety. Red Blood Cell Count detects the effect of Sanggua tablets on the number of red blood cells, determine whether there is anemia or increased red blood cells, and evaluate the effect of Sanggua tablets on hematopoietic function. Evaluate whether these indicators are within the normal range during the treatment period.
Hemoglobin (Hb, g/L) | Hemoglobin will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Blood routine examination is a standard test that evaluates the levels of red and white blood cells, platelets, and other components in the blood, providing a general overview of health and the tablets' safety. Hemoglobin evaluates the impact of Sanggua tablets on hemoglobin levels, determine whether there is anemia or abnormal hemoglobin, and reflect the effect of Sanggua tablets on oxygen transport capacity. Evaluate whether these indicators are within the normal range during the treatment period.
Platelet Count (PLT, 10^9/L) | Platelet Count will be measured at the following time points during the clinical trial: enrollment visit (V1), Week 4 (V2), and Week 16 (V5).
  Blood routine examination is a standard test that evaluates the levels of red and white blood cells, platelets, and other components in the blood, providing a general overview of health and the tablets' safety. Platelet Count detects the effect of Sanggua tablets on the platelet count, determine whether there is thrombocytopenia or thrombocytopenia, and evaluate the effect of Sanggua tablets on coagulation function and bleeding risk. Evaluate whether these indicators are within the normal range during the treatment period.
diabetes self-care activities scale(SDSCA) | Participants will complete the SDSCA at baseline (V1) and at the end of the treatment period(Week 16 ,V5).
  We will use summary of diabetes self-care activities scale(SDSCA) to evaluate and standardize participants' lifestyle factors, ensuring that the observed effects on glycemic control can be accurately attributed to the treatment rather than dietary or exercise changes. The Likert 8-level scoring system is adopted, with a total score ranging from 0 to 77 points. The higher the score, the better the self-management behavior. Evaluate whether the scale scores are within the similar range during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Yuan, Professor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China